CLINICAL TRIAL: NCT04139187
Title: Lower Extremities Biomechanics Responses to Power and Strength Combined Training in Adults: a Randomized Clinical Trial
Brief Title: Biomechanics Responses to Power and Strength Combined Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Collaborators: Universidade Federal do Pampa (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Karine Josibel Velasques Stoelben, Principal Investigator, Universidade Federal do Pampa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96793518.3.0000.5323
Record Dates: First submitted 2019-09-04; First posted 2019-10-25 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Adult; Anterior Cruciate Ligament Injuries; Lower Extremity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Two groups design where one randomized group receive treatment and the other not in the same period of time.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistical analyzer will be masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Individuals randomized to experimental group.
  Interventions: Other: Combined training with power and strength exercises
- No Intervention Control (No Intervention): Individuals without quadriceps dominance randomized to no intervention group.

INTERVENTIONS:
Other: Combined training with power and strength exercises — The training will be compose by power and strength exercises and divided in two days. One day with the exercises: vertical jumps, box jumps, sit-ups, back-extension and guided squat. The second with half squat jumps, high straight jumps, bounding jumps, drop jumps and sprint. Both days will be started with warm up on treadmill running lasting 5 minutes at 6.5-7.5 km/h.
  The training protocol includes 20 sessions with 2 sessions per week during 10 weeks (2 weeks to adaptation and others 8 to training with progression of load after 4 weeks).
  Arms: Experimental

SUMMARY:
Anterior cruciate ligament (ACL) is the most frequently injured knee ligament during performance of recreational activities and sports. In the United States, the annual incidence is 68.6 per 100,000 people per year and in Brazil, the estimation of ACL reconstruction increases 64%. There are different biomechanical profiles of risk factors for an ACL injury variable, the ligament dominance, the quadriceps dominance, the trunk dominance, and the leg dominance. Thus, the purpose of this study is to investigate the biomechanics adaptations after power and strength combined training protocol in healthy individuals. A second aim is to determine the effect of the training on knee injury risk factors.

DETAILED DESCRIPTION:
This is a parallel randomized clinical trial comparing the effect of combined training with power and strength exercises on lower extremity biomechanics in healthy individuals.

The sample size was calculated with G*Power software using the ANOVA: Repeated measures, within-between interaction, 90% power, alpha 0.05, and 30% drop-out. Data from the tuck jump test (knee flexion range) by Makaruk (2014) were considered for this calculation with effect size 0.46. Thus, a total of 32 individuals (16 per group) is required for this study. To ensure the proper simple size, after collecting the first five participants per group, the sample size will be checked again.

The participants will be randomized in experimental and no intervention groups inside each risk profile group. Randomization ratio will be 1:1 and interventions will last 10 weeks, with two weekly sessions for the exercise arms.

The outcomes will include functional clinical tests, kinematic and kinetic variables during landing tasks, and strength of knee and hip muscles.

The data analysis will be performed by intention to treat and per protocol. Generalized estimating equations will be used to identify interaction effects of groups and time followed by Bonferroni post-hoc. When effect are found, effect size will be estimated. Missing data will be estimate by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male sex;
* Age between 18 and 30 years old;
* Who practice physical activity (except: strength and jump training) between 80 and 150 minute per week;
* No previous muscle lower extremity injury at least 6 months prior to recruitment;
* No previous ligament and tendon lower extremity injury or surgery;
* No auditory, vestibular, visual or musculoskeletal injuries or disease that impairment the execution of assessments or training protocol;
* No hypertension, cardiovascular or respiratory disease.

Exclusion Criteria:

* Body mass index greater than 35 kg/m².

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline peak sagittal plane angle of ankle, knee and hip from both legs | Baseline and up to 10 weeks
  Peak angle of sagittal plane during landing task
Change from baseline value of sagittal plane angles for ankle, knee, hip, pelvis from both legs, and trunk | Baseline and up to 10 weeks
  Value at initial contact instant and maximal knee flexion instant of landing task
Change from baseline value of frontal plane angles for ankle, knee, hip, pelvis from both legs, and trunk | Baseline and up to 10 weeks
  Value at initial contact instant and maximal knee flexion instant of landing task
Change from baseline value of transverse plane angles for hip, pelvis from both legs, and trunk | Baseline and up to 10 weeks
  Value at initial contact instant and maximal knee flexion instant of landing task
Change from baseline peak frontal plane angle of knee and hip from both legs | Baseline and up to 10 weeks
  Peak angle of frontal plane during landing task
Change from baseline range of knee frontal plane angle from both legs | Baseline and up to 10 weeks
  Range of frontal plane angle between initial contact instant and maximal knee flexion instant of landing task
Change from baseline range of knee sagittal plane angle from both legs | Baseline and up to 10 weeks
  Range of sagittal plane angle between initial contact instant and maximal knee flexion instant of landing task
Change from baseline value of sagittal plane joint moment knee and hip from both legs | Baseline and up to 10 weeks
  Value at initial contact instant and maximal knee flexion instant of landing task
Change from baseline value of frontal plane joint moment knee and hip from both legs | Baseline and up to 10 weeks
  Value at initial contact instant and maximal knee flexion instant of landing task
Change from baseline peak of knee frontal plane joint moment from both legs | Baseline and up to 10 weeks
  Peak of joint moment during landing task
Change from baseline value of ground reaction force vertical component from both legs | Baseline and up to 10 weeks
  Value at maximal knee flexion instant of landing task
Change from baseline value of loading rate from both legs | Baseline and up to 10 weeks
  Value calculated by relation between peak of ground reaction force vertical component and time to peak from initial contact during landing task
Change from baseline peak of ground reaction force vertical component from both legs | Baseline and up to 10 weeks
  Peak of ground reaction force during landing task
Change from baseline value of muscle maximal isometric strength for knee extensors and flexors, and hip aductors and abductors from both legs | Baseline and up to 10 weeks
  Value of maximal isometric strength

SECONDARY OUTCOMES:
Change from baseline pennation angle of muscle fibers of knee extensors and flexors from both legs | Baseline and up to 10 weeks
  The angle between the longitudinal axis of the entire muscle and its fibers.
Change from baseline muscle fascicle length of knee extensors and flexors from both legs | Baseline and up to 10 weeks
  The distance between the intersection composed of the superficial aponeurosis and fascicle and the intersection composed of the deep aponeurosis and the fascicle
Change from baseline muscle thickness of knee extensors and flexors from both legs | Baseline and up to 10 weeks
  Estimation of muscle cross-sectional area
Change from baseline power value of ankle, knee and hip joints from both legs | Baseline and up to 10 weeks
  Relation of work and velocity during landing task
Change from baseline dynamic strength of lower extremities muscles | Baseline and up to 10 weeks
  The force developed to perform one maximal repetition to perform leg press and squat tasks
Change from baseline maximal dorsiflexion amplitude of ankle joint from both legs | Baseline and up to 10 weeks
  Maximal dorsiflexion amplitude obtained during lunge test
Change from baseline dynamic balance of lower extremities from both legs | Baseline and up to 10 weeks
  Dynamic balance is assessed according the displacement obtained during Star Excursion Balance Test
Change from baseline dynamic balance index of asymmetry between legs | Baseline and up to 10 weeks
  Dynamic balance is assessed according the displacement obtained during Star Excursion Balance Test. The asymmetry index is calculated by relation between preferred and non preferred legs.
Change from baseline quality of dynamic movement of lower extremities from both legs | Baseline and up to 10 weeks
  Quality of movement is assessed according the escore obtained during Lateral Step Down test performance
Change from baseline asymmetry index of quality of dynamic movement between legs | Baseline and up to 10 weeks
  Quality of movement is assessed according the escore obtained during Lateral Step Down test performance. The asymmetry index is calculated by relation between preferred and non preferred legs.
Change from baseline functional physical performance of lower extremities from both legs | Baseline and up to 10 weeks
  Assessed according the maximal distance obtained during hop tests performance (single, triple and crossover)
Change from baseline asymmetry index of functional physical performance between legs | Baseline and up to 10 weeks
  Assessed according the maximal distance obtained during hop tests performance (single, triple and crossover). The asymmetry index is calculated by relation between preferred and non preferred legs.

OTHER OUTCOMES:
Training load of each training session | At the end of each training session throughout 10 weeks
  Product between rate of perceived exertion and session duration training
Muscle Soreness after each training session | 24 and 48 hours after each training session throughout 10 weeks
  Value from visual analog scale (score between 0 to 10 points) representative to discomfort or pain after training sessions. Higher values represent worst discomfor/pain

CONTACTS AND LOCATIONS:
Overall Officials: Felipe P Carpes, PhD, Study Director — Federal University of Pampa; Karine JV Stoelben, Ms, Principal Investigator — Federal University of Pampa; Eliane C Guadagnin, PhD, Study Chair — Federal University of Pampa
Locations (1):
- Karine Josibel Velasques Stoelben, Uruguaiana, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to publish the results in an open-access journal, indexed at the Directory of Open Access Journals, with the copyrights transferred to the authors. Details regarding the study's design and statistical plan can be obtained consulting the trial's protocol. Data on other outcomes could be requested contacting the PI.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The individual participant dataset will become available at a public repository up to six months after the first study publication
Access Criteria: A simple registration will grant access to study datasets. The website for these files is not defined at the time of registration.